CLINICAL TRIAL: NCT03937583
Title: PET / CT Scan to Detect Cancer in Patients With Unprovoked Venous Thromboembolic Disease. Open Randomized Clinical Trial.
Brief Title: Screening for Cancer in Patients With Unprovoked VTE
Acronym: SOME-RIETE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: SOME RIETE; 2018-003958-25 (EudraCT Number)
Record Dates: First submitted 2019-04-30; First posted 2019-05-06 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: Venous Thromboembolic Disease; Respiratory Disease; Pulmonary Disease; Deep Venous Thrombosis; Pulmonary Embolism; Screening; Undefined
Keywords: Venous Thromboembolic Disease; Pulmonary Embolism; Screening; Occult Cancer
MeSH Terms: conditions — Respiration Disorders; Lung Diseases; Venous Thrombosis; Pulmonary Embolism | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited screening (No Intervention): Complete clinical history, along with routine physical, analytical examination (creatinine, sodium, potassium, red series, white series, liver and calcium profile) and chest x-ray.
- Extended screening (Experimental): Limited screening plus positron emission tomography / computed tomography with 18 FDG (18FDG PET-CT).
  Interventions: Drug: Fludeoxyglucose 18F

INTERVENTIONS:
Drug: Fludeoxyglucose 18F — The performance of the 18 FDG PET-CT will require fasting of at least 6 hours, and the glycemia will have to be lower than 126 mg / dL before the injection of 3-5 MBq / kg of 18FDG. Intravenous injection will follow a period of approximately 60 minutes in a quiet room.
  Computed tomography (CT) will be performed from the middle of the forehead to the feet with normal and shallow breathing using a low dose adjustment Iodinated contrast will not be administered intravenously.
  Other Names: 18-Fludeoxyglucose (18FDG)
  Arms: Extended screening

SUMMARY:
Open and multicenter randomized clinical trial (1:1) comparing limited screening with extended screening with the performance of Positron emission tomography-computed tomography (PET-CT) scan in the search for neoplasms in patients with unprovoked venous thromboembolic disease at high risk of developing cancer at follow-up.

Introduction: Cancer screening in patients with unprovoked venous thromboembolic disease (VTE) is controversial. In the last years, a score has been developed that selects patients at high risk of developing cancer during follow-up.

Objective: To estimate the impact of an active cancer search strategy using 18-fluordesoxiglucose (FDG) PET-CT in unprovoked VTE with high-risk to develop cancer.

Specific Objectives: 1) Number of neoplasms diagnosed in the screening process: 2) number of neoplasms diagnosed at an early stage, 3) impact on survival of the strategy; and 4) impact on the quality of life.

Cancer will be considered from 30 days up to 12 months after the diagnosis of VTE.

Scope: 20 Spanish hospitals. Design: Open-label, multicentre Randomized clinical trial (1: 1) comparing the performance of PET-CT versus limited screening for cancer.

Population: Patients older than 18 years with unprovoked VTE at high risk of presenting cancer at follow-up (≥3 points in the score of Jara-Palomares et al., Chest 2017).

Follow-up: 12 months after VTE. Sample: The sample size calculated is 650 patients, to obtain a power of 80%, with a level of significance of 5%, and taking into account a 10% loss of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* Diagnosis of venous thromboembolic disease (proximal deep vein thrombosis of lower limbs, pulmonary embolism or both) unprovoked.
* High risk classification according to previously published and validated scale
* Signature of informed consent form

Exclusion Criteria:

* Impossibility to continue an adequate follow-up.
* Contrast hypersensitivity used for PET / CT (fludeoxyglucose (18FDG)) or any of the excipients according to the characteristics of the product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2019-10-23 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of neoplasms diagnosed using extended screening | After 3 years of follow-up
  Estimate the impact of an active cancer search strategy using PET-CT in the number of neoplasms diagnosed in the screening process in patients with high-risk unprovoked thromboembolic disease.

SECONDARY OUTCOMES:
Number of neoplasms diagnosed in early phase using extended screening | After 3 years of follow-up
  Estimate the impact of an active cancer search strategy using PET-CT in the number of neoplasms diagnosed in early phase in the screening process in patients with high-risk unprovoked thromboembolic disease.
Overall survival of patients with high-risk unprovoked thromboembolic disease performing limited/extended screening | Until the patient death or finalization of study after three years of follow-up
  Estimate the impact of an active cancer search strategy using PET-CT in the overall survival in patients with high-risk unprovoked thromboembolic disease.
European Quality of Life-5 (EQ-5D scale validated in Spanish) of patients with high-risk unprovoked thromboembolic disease performing limited/extended screening | Baseline and after 90, 180 and 365 days of follow-up
  Estimate the impact of an active cancer search strategy using PET-CT in the quality of life evaluated with the scale EQ-5D in patients with high-risk unprovoked thromboembolic disease. The EQ-5D consists of 2 parts - the "Descriptive System" and the "Visual Analogue scale". The DS comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems.
  The EQ VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Jara Palomares, MD/PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío
Locations (17):
- Spain (17):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Fundació Hospital de L'Esperit Sant, Santa Coloma de Gramenet, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville, Seville
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d'Hebrón, Barcelona
  - Consorcio Hospitalario Provincial de Castellón, Castelló
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital de Granollers, Granollers
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Infanta Sofía, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clínica Universidad de Navarra, Pamplona
  - Hospital Universitario de Valme, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD to be shared with the center participants once the study is officially finished in the foreseen period of three years.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 3 years time
Access Criteria: In order to access the data, the study must first be completed, the database must be closed, and analyzed. Once the manuscript is written, the results will be sent to the participating centers, and study data may be requested upon request to the principal investigator who will evaluate together with the study investigators.

REFERENCES:
- [Derived] Barca-Hernando M, Otalora-Valderrama S, Lopez-Nunez JJ, Portillo-Sanchez J, Pagan-Escribano J, Lopez-Miguel P, Mahe I, Mena-Munoz E, Jou-Segovia I, Imbalzano E, Agudo-de Blas P, Lorenzo-Hernandez A, Diaz-Pedroche C, Aibar-Gallizo J, de la Red-Bellvis G, Del Molino-Sanz F, Amado-Fernandez C, Fernandez-Reyes JL, Villalobos-Sanchez A, Lopez-Saez JB, Diaz-Brasero AM, Marcos-Jubilar M, Meireles J, Marchena-Yglesias PJ, Diaz-Peromingo JA, Marin-Romero S, Elias-Hernandez T, Andrade-Ruiz HA, Mehdipour G, Bikdeli B, Jara-Palomares L; SOME-RIETE and ValRIETEs Investigators. Occult cancer in patients with unprovoked venous thromboembolism: Rationale, design, and methods of the VaLRIETEs study and the SOME-RIETE trial. Am Heart J. 2025 Jun;284:81-93. doi: 10.1016/j.ahj.2025.02.004. Epub 2025 Feb 17. PMID 39971173